CLINICAL TRIAL: NCT05007002
Title: Robot-based Therapy for Upper Limb Sensorimotor Impairments in the Chronic Phase After Stroke: a Pilot Study
Brief Title: Robot-based Therapy for Upper Limb Sensorimotor Impairments After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Professor Neurorehabilitation, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S61997[2]
Record Dates: First submitted 2021-07-11; First posted 2021-08-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Somatosensation; Sensory processing; Proprioception; Robot-based therapy; Robot-based assessment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-based therapy (Experimental): Chronic stroke patients receiving robot-based therapy
  Interventions: Device: Robot-based therapy

INTERVENTIONS:
Device: Robot-based therapy — Active and passive therapy tasks for proprioception and sensory processing, with use of the Kinarm End-Point Lab (BKIN Technologies Ltd., Canada)

SUMMARY:
After a stroke, more than two out of three patients experience problems with upper limb movement and sensation. Current evidence on treatment of upper limb sensory impairments is scarce and shows unclear results. Robot-based therapy has been increasingly used to treat upper limb motor impairments, with similar positive results as compared to conventional therapy. This study aims to investigate a novel robot-based therapy program for treatment of upper limb sensory impairments. The therapy program consists of 10 one-hour session spread over 4 weeks and will be evaluated for its effect in 20 chronic stroke patients. The investigators hypothesize that a 4-week robot-based therapy program can improve upper limb sensation and movement.

DETAILED DESCRIPTION:
Up to 70% of stroke survivors show upper limb impairments consisting of motor and/or somatosensory impairments. These impairments often persist well into the chronic stage, and may lead to significant limitations in activities of daily living and may negatively affect quality of life. Different interventions have been investigated to treat upper limb motor impairments, including robot-based therapy, which shows similar positive results as compared to conventional therapy. Evidence on interventions for somatosensory impairments is scarce and often of low quality. This study therefore aims to evaluate the effect of a robot-based therapy program on sensorimotor function of the upper limb in a group of 20 chronic stroke patients.

The robot-based therapy will be provided using the Kinarm End-Point Lab (BKIN Technologies Ltd., Canada) and consists of passive and active therapy tasks for proprioception and sensory processing. The therapy consists of 10 one-hour sessions spread over 4 weeks. Clinical and robot-based motor and somatosensory assessments will be performed at 4 time points: twice at baseline, once at mid intervention, and once after 10 hours of therapy. The investigators hypothesize to find improvement in both upper limb motor and somatosensory function after the therapy program. The results from this pilot study will provide a basis for further research.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* A first-ever unilateral, supratentorial stroke (as defined by WHO)
* In the chronic phase after stroke (i.e. being at least 6 months after stroke)
* Motor deficits of the upper limb (Fugl-Meyer Motor Assessment - Upper Extremity < 60/66)
* Somatosensory deficits of the upper limb (Erasmus modified Nottingham Sensory Assessment < 36/40)
* Ability to perform, at least to some extent, active shoulder abduction and wrist extension against gravity
* Ability to perform passive and active sensory processing assessment task (primary outcome measure)

Exclusion Criteria:

* History of previous stroke or TIA
* Any serious musculoskeletal and/or other neurological conditions
* Serious communication or cognitive deficits
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Kinarm: sensory processing task | Change during 4 weeks of therapy provided at least 6 months after stroke
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing

SECONDARY OUTCOMES:
Kinarm: arm position matching task | Change during 4 weeks of therapy provided at least 6 months after stroke
  Assessment of limb position sense using a 9-target mirror-matching task on the Kinarm Exoskeleton Lab
Kinarm: arm movement matching task | Change during 4 weeks of therapy provided at least 6 months after stroke
  Assessment of limb movement sense using a mirror-matching task on the Kinarm Exoskeleton Lab
Kinarm: visually guided reaching task | Change during 4 weeks of therapy provided at least 6 months after stroke
  Assessment of motor function using a 4-target centre-out reaching task on the Kinarm End-Point Lab
Kinarm: working memory task | Change during 4 weeks of therapy provided at least 6 months after stroke
  Assessment of working memory on the Kinarm End-Point Lab, by asking the participant to remember the position of 3, 4, 5 or 6 targets simultaneously.
Erasmus modified Nottingham sensory assessment | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of somatosensory function (including exteroception, proprioception and sensory processing) on an ordinal scale ranging from 0 to 40, with higher scores meaning better performance
Tactile discrimination test | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Functional tactile object recognition test | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 42, with higher scores meaning better performance
Fugl-Meyer upper extremity assessment | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of motor function on an ordinal scale ranging from 0 to 66, with higher scores meaning better performance
Action research arm test | Change during 4 weeks of therapy provided at least 6 months after stroke
  Timed clinical assessment of motor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Sensorimotor action research arm test | Change during 4 weeks of therapy provided at least 6 months after stroke
  Timed clinical assessment of sensorimotor performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Montreal cognitive assessment | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of cognitive function on an ordinal scale ranging from 0 to 30, with higher scores meaning better performance
Star cancellation test | Change during 4 weeks of therapy provided at least 6 months after stroke
  Clinical assessment of visuospatial neglect on an ordinal scale ranging from 0 to 54, with higher scores meaning better performance, and a score below 44 indicating the presence of visuospatial neglect
Kinarm: sensory processing task | Change in 2 baseline measures taken 2 days apart, at least 6 months after stroke
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing
Kinarm: sensory processing task | Change during the first 2 weeks of a 4-week therapy protocol provided at least 6 months after stroke
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing
Kinarm: sensory processing task | Change during the last 2 weeks of a 4-week therapy protocol provided at least 6 months after stroke
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided